CLINICAL TRIAL: NCT03034148
Title: Prospective Evaluation of Acetyl-Coenzyme A Carboxylase Phosphorylation State in Platelets in Atherothrombotic Coronary Artery Disease.
Brief Title: Platelet Acetyl Coenzyme A Carboxylase Phosphorylation in Coronary Artery Disease
Acronym: ACCTHEROMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: cb07012015
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; Coronary Thrombosis
Keywords: Coronary artery disease; Atherothrombosis; Thrombin generation; Platelet Acetyl Coenzyme A carboxylase phosphorylation
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Coronary Thrombosis; Thrombosis | interventions — Diagnosis, Computer-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Coronary artery disease (Other): blood sampling for biomarkers assessment in a population undergoing coronary angiogram
  Interventions: Diagnostic Test: Platelet Acetyl Coenzyme A Carboxylase analysis in CAD

INTERVENTIONS:
Diagnostic Test: Platelet Acetyl Coenzyme A Carboxylase analysis in CAD

SUMMARY:
In human purified platelets, only thrombin, and not the other platelet agonists, leads to a transient activation of the protein kinase activated by AMP (AMPK) and to phosphorylation of its "bona fide" substrate, ACC on its Ser79. ACC phosphorylation (P-ACC) can be an interesting marker of thrombin action on platelets. Indeed platelet and coagulation interplay, though undoubtedly present in atherosclerosis and atherothrombosis, remains difficult to assess. Our group showed that atherosclerotic mice (SRBI/Apolipoprotein E knock-out) had higher platelet P-ACC compared to corresponding control mice (C57BL6). In agreement with these data, preliminary results showed increased platelet P-ACC in a small cohort of patients admitted for coronary angiogram, with demonstrated coronary artery disease (CAD).

In the light of our preliminary results, we sought to analyze platelet P-ACC in a large prospective clinical trial (ACCTHEROMA) in patients admitted for coronary angiogram. The aim of the study is to compare platelet P-ACC in platelets of patients with CAD and more particularly in unstable CAD patients to non-CAD patients. This study could potentially identify patients at high risk of future ischemic cardiovascular events, because of a higher level of thrombin generation.

DETAILED DESCRIPTION:
Consecutive patients with planned coronary angiogram at the Cliniques Universitaires Saint Luc, Brussels, whatever the indication, will be included between March 2015 and February 2016. Informed consent will be obtained before angiogram.

A. Blood Sampling Routine veinous blood sample will be done under fasting condition in the cardiology ward before the angiogram (standard of care for patients undergoing coronary angiogram).

In order to avoid additional puncture for blood sampling and to limit platelet activation, blood samples are withdrawn after sheath insertion at the Cath lab before any drug administration. The following measurements will be done:

* Routine coagulation tests including international rationalize ratio, activated cephaline time, thrombin time, prothrombin time, Fibrinogen, DDimers.
* Platelet reactivity testing by the Multiple Electrode Aggregometer (Multiplate Analysis)
* Platelet isolation and lysates will be stocked frozen for phospho-protein analysis by immunoblotting and electrochemiluminescence (ECLIA)
* Aliquots of poor platelet plasma stocked frozen for inflammation (HsCRP), thrombin generation tests (thrombin-antithrombin complex, prothrombin fragment F1.2, endogenous thrombin generation potential-ETP), platelet activation markers (platelet factor 4, soluble CD40ligand, soluble P-selectin) and circulating micro-RNA extraction.
* Platelet isolation and further purification for platelet specific micro-RNA extraction.

B. Atherosclerosis evaluation All patients underwent coronary angiogram. Significant coronary artery lesion is defined as a luminal stenosis above 50%. Syntax score will be calculated for all patients.

Global atherosclerotic plaque burden on coronary and extracoronary arteries will be evaluated by measuring calcium score on thoraco-abdominal scanner with prospective ECG-gating in a randomly selected subgroup of patients. Coronary artery calcification (CAC) is expressed as Agatston score using calcium scoring software (Philips Healthcare) with a threshold of 130 Hounsfield units. The degree of atherosclerotic burden on coronary arteries is classified as mild (Agatston score <100), moderate (Agatston score 100-400) or severe (Agatston score >400). Aortic calcification (AoC score) was measured from aortic arch to iliac arteries in all patients.

C. Data collection Baseline characteristics of patients will be collected from the medical database of the Cliniques Universitaires Saint Luc. All coronary angiogram will be reviewed by 2 different investigators and syntax score will be calculated with the online syntax score calculator. CAC Agatston and AoC score will also be assessed by 2 different investigators.

D.Patients Classification for platelet P-ACC analysis Platelet ACC phosphorylation (P-ACC) analysis will be done by immunoblotting with a specific antibody probing for phosphorylated (Ser 79) ACC. Purified washed platelets stimulated with 0.5 units/ml thrombin will be used as positive internal controls.

Patients will first be classified in non-CAD and CAD groups based on the results of coronary angiogram and CAC Agatston score: Non-CAD (absence of lesion on angiogram and/or CAC Agatston score<100) and CAD (presence of at least 1 lesion on angiogram and/or CAC Agatston score>100).

In a second analysis, based on clinical presentation, the CAD group will further be divided into Stable CAD or Unstable CAD [acute coronary syndrome (ACS)]. Platelet P-ACC will be compared in both subgroups. This detailed classification will outline high-risk patients with ongoing acute coronary syndrome.

E. Sample size and statistical analysis. Based on our preliminary data, we determined that enrolment of 102 patients would provide a power of 80% at a significance level of 5% to detect a difference of 0.15 (A.U.) in the phosphorylation of ACC in atherosclerotic patients, compared to non CAD patients.

Continuous variables will be expressed as mean +/- one standard deviation, categoric variables as counts and percentages. Patients will separated in four groups depending on the level of P-ACC (quartiles). Clinical presentation, thrombin generation markers and calcium scoring will be compared in all these groups, based on ANOVA analysis. Variables will be submitted to logistic regression test in order to identify independent predictors of high ACC phosphorylation state. The role of high platelets P-ACC in assessing the risk of the patients will be then studied.

F.Follow-up A follow-up period of 3 years is planned. Events recorded during the follow-up period will be obtained from the medical database and a phone call will be done in case of missing data.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Planned angiography within the next 3 days, whatever the indication.

Exclusion Criteria:

* Not able to sign informed consent
* Patients on anticoagulation therapy (oral or parenteral) including heparins, fondaparinux, vitamin K antagonist, novel oral anticoagulants, for any reasons.
* Active neoplasia
* Active inflammatory disease
* Patients with life expectancy lower than 3 years
* Haemophilia and other coagulopathy
* Abnormal platelet count
* Heart transplanted patients
* Active hepatitis B or C or HIV patients
* Any contra-indication for coronary angiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
an increase in platelet ACC phosphorylation state in patients with coronary artery disease | 2 years

SECONDARY OUTCOMES:
a correlation between thrombin generation markers and platelet P-ACC in overall population. | 2 years
platelet ACC phosphorylation state according clinical severity of CAD (stable versus unstable patients) | 2 years
the role of platelet P-ACC in predicting the risk of the patient for future cardiovascular events (death, myocardial infarction, stroke) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Beauloye, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Onselaer MB, Oury C, Hunter RW, Eeckhoudt S, Barile N, Lecut C, Morel N, Viollet B, Jacquet LM, Bertrand L, Sakamoto K, Vanoverschelde JL, Beauloye C, Horman S. The Ca(2+) /calmodulin-dependent kinase kinase beta-AMP-activated protein kinase-alpha1 pathway regulates phosphorylation of cytoskeletal targets in thrombin-stimulated human platelets. J Thromb Haemost. 2014 Jun;12(6):973-86. doi: 10.1111/jth.12568. PMID 24655923
- [Derived] Robaux V, Kautbally S, Ginion A, Dechamps M, Lejeune S, Menghoum N, Bertrand L, Pouleur AC, Horman S, Beauloye C. Dual antiplatelet therapy is associated with high alpha-tubulin acetylation in circulating platelets from coronary artery disease patients. Platelets. 2023 Dec;34(1):2250002. doi: 10.1080/09537104.2023.2250002. PMID 37700239